CLINICAL TRIAL: NCT07305623
Title: Phase III Randomized Clinical Trial on the Use of a Bone Bioengineering Kit With Stem Cells Versus Autogenous Iliac Crest Graft for Alveolar Cleft Repair in Patients With Cleft Lip and Palate
Brief Title: Safety and Efficacy of Bone Bioengineering Kit With Stem Cells for Alveolar Cleft Repair
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Tecnologia do Paraná (Other)
Responsible Party: Principal Investigator, Daniela Franco Bueno, DDS, PhD, Instituto de Tecnologia do Paraná
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TECPAR_2025
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cleft Lip Palate
Keywords: bioengineering kit; Stem cells
MeSH Terms: interventions — Biocompatible Materials

STUDY DESIGN:
Intervention Model Description: Patients will receive the bioengineering kit composed of stem cells from deciduous teeth and biomaterial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioengineering kit (Experimental): Patients will receive the bioengineering kit composed of stem cells from deciduous teeth and biomaterial.
  Interventions: Combination Product: Bioengineering kit composed of stem cells from deciduous teeth and biomaterial.
- Iliac crest bone graft (Active Comparator): Standard iliac crest bone graft surgery
  Interventions: Procedure: iliac crest bone graft surgery

INTERVENTIONS:
Combination Product: Bioengineering kit composed of stem cells from deciduous teeth and biomaterial. — Bone tissue engineering kit composed of 10⁶ mesenchymal stromal cells/mesenchymal stem cells (MSCs) derived from dental pulp, combined with a biomaterial consisting of hydroxyapatite and collagen (BioOss Collagen, 250 mg, Geistlich).
  Arms: bioengineering kit
Procedure: iliac crest bone graft surgery — standard iliac crest bone graft surgery
  Arms: Iliac crest bone graft

SUMMARY:
The objective of this study is to compare the safety and efficacy of the bone tissue engineering kit-composed of 10⁶ mesenchymal stem cells derived from deciduous dental pulp combined with a collagen- and hydroxyapatite-based biomaterial-with secondary autogenous bone grafting for alveolar cleft closure in patients with cleft lip and palate.

Individuals aged 6 to 11 years with unilateral pre- and transforamen cleft lip and palate who have an indication for bone grafting will be included.

The study will be conducted in two stages. In Stage 1, patients will undergo surgery using only the bioengineering kit, and the primary outcome will be the average length of hospital stay after grafting with the engineering kit. In Stage 2, patients will be randomized to receive either the bioengineering kit treatment or the standard iliac crest bone graft surgery. In this stage, the primary outcome will be the success rate of the cleft lip and palate repair surgery, determined by the amount of bone formation in the alveolar cleft region, measured through volumetric analyses of computed tomography scans performed 12 months after grafting.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (ICF) from the legal guardian;
* Signed Assent Form from the participant;
* Patients aged 6 to 11 years at the time of the secondary bone graft surgery;
* Participants diagnosed with unilateral cleft lip and palate of the pre-foramen incisive or transforamen type;
* Patients must have had mesenchymal stem cells derived from deciduous teeth collected and stored in a biobank prior to signing the Informed Consent Form (ICF);
* Patients with the maxilla previously aligned through orthodontic treatment and deemed suitable for the alveolar bone graft procedure;
* Patients who are reliable and willing to be available throughout the study, attend all required study visits, and are willing and able to comply with study procedures as necessary.

Exclusion Criteria:

* Previous surgery for alveolar cleft repair;
* Presence of comorbidities (diabetes, cardiac conditions, hypertension) or allergies to latex gloves and suture materials (Catgut, Vicryl, Monocryl, Nylon, Polyester, or Polypropylene);
* Presence of palatal fistulas resulting from previous surgeries;
* Incomplete orthodontic or tomography documentation;
* Eruption of the permanent canine prior to signing the Informed Consent Form (ICF) and Assent Form (AF), and prior to undergoing the secondary alveolar bone graft surgery;
* Participants who are pregnant or breastfeeding at the time of screening or during the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 205 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of the cleft lip and palate repair surgery | 12 months
  average amount of bone formation in the alveolar cleft region, measured through volumetric analyses of computed tomography scans

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pequeno Príncipe, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No